CLINICAL TRIAL: NCT00895089
Title: Prospective, Randomized, Open-Labeled, Active-Controlled Comparison of Moxifloxacin Versus Ceftriaxone in the Treatment of Primary Pyogenic Liver Abscess: A Pilot Study
Brief Title: Moxifloxacin Versus Ceftriaxone in the Treatment of Primary Pyogenic Liver Abscess
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Susan Shin-Jung Lee, Attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS98-CT2-20
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Liver Abscess
Keywords: liver abscess; moxifloxacin; ceftriaxone; treatment
MeSH Terms: conditions — Liver Abscess | interventions — Moxifloxacin; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Moxifloxacin (Experimental): Moxifloxacin 400mg IV once daily for 14 days, then 400mg PO once daily for 7 days.
  Interventions: Drug: Moxifloxacin (Avelox)
- B: Ceftriaxone (Active Comparator): Ceftriaxone 2gm IV every 12 hours for 14 days, then cephalexin 1gm PO every 6 hours for 7 days.
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: Moxifloxacin (Avelox) — moxifloxacin 400 mg IV qd for 14 days, followed by moxifloxacin 400 mg po qd for another 1 week
  Other Names: Avelox
  Arms: A: Moxifloxacin
Drug: ceftriaxone — ceftriaxone 2 gm IV q 12 h for 14 days, followed by cephalexin 1 gm PO q 6 h for 1 week
  Other Names: Rocephin; Cefin
  Arms: B: Ceftriaxone

SUMMARY:
This clinical trial compares the use of moxifloxacin versus ceftriaxone in the treatment of primary pyogenic liver abscess. The trial will include nonpregnant adults presenting with primary liver abscess based on clinical diagnosis and computed tomography. The trial aims to determine whether the use of moxifloxacin can effectively treat primary pyogenic liver abscess and shorten hospitalization. This regimen has the additional benefit of avoiding nephrotoxic agents, such as aminoglycosides, used frequently in treatment of pyogenic liver abscess. Development of antibiotic resistance to colonized bacteria in the gastrointestinal tract will also be evaluated using stool cultures.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 20 years.
* Clinical diagnosis of liver abscess, supported by an abdominal CT scan, documenting the presence of liver abscess, in the absence of biliary tract stones (except for gallstones without biliary tract dilatation), biliary tract dilatation and biliary tract tumors. Clinical diagnosis of liver abscess includes symptoms of fever, chills, right upper quadrant abdominal pain or knocking tenderness.
* Read, understood and signed informed consent form.

Exclusion Criteria:

* Presence of septic metastatic infections to the CNS or eye at presentation.
* Cultures positive for an organism resistant to study drugs.
* APACHE II score greater or equal to 20.
* Co-existent disease considered likely to affect the outcome of the study (e.g., biliary tract stones and malignancy).
* Patients with ruptured liver abscess
* Severe hepatic insufficiency (Child-Pugh C) or elevated serum transaminases (GPT) to greater than 5 times the upper limit of normal.
* Patients who are pregnant or lactating.
* Known hypersensitivity to b-lactams or fluoroquinolones.
* Known prolongation of the QT interval.
* Patients with uncorrected hypokalemia.
* Patients receiving class IA (e.g., quinidine, procainamide) or class III (e.g., amiodarone, sotalol) antiarrhythmic agents
* Severe, life-threatening disease with a life expectancy of less than 2 months.
* Pre-treatment with a systemic antibacterial agent for > 24 hours prior to enrollment within 5 days prior to enrollment.
* Participated in any clinical investigational drug study within 4 weeks of screening.
* Previously entered in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | 21 days

SECONDARY OUTCOMES:
Clinical response | Day 3, 7 and 14
Clinical and radiological response | 21 days
All cause mortality | 21 days
Mortality attributable to liver abscess during treatment | 21 days
Rates of complication (metastatic infections to the central nervous system and/or eyes) | 21 days
Rates of gastrointestinal colonization of Klebsiella pneumoniae in patients and rates of resistance post-antibiotic use. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shin-Jung Lee, M.D., M.Sc, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lee SS, Chen YS, Tsai HC, Wann SR, Lin HH, Huang CK, Liu YC. Predictors of septic metastatic infection and mortality among patients with Klebsiella pneumoniae liver abscess. Clin Infect Dis. 2008 Sep 1;47(5):642-50. doi: 10.1086/590932. PMID 18643760
- [Background] Tsai FC, Huang YT, Chang LY, Wang JT. Pyogenic liver abscess as endemic disease, Taiwan. Emerg Infect Dis. 2008 Oct;14(10):1592-600. doi: 10.3201/eid1410.071254. PMID 18826824
- [Background] Liu YC, Cheng DL, Lin CL. Klebsiella pneumoniae liver abscess associated with septic endophthalmitis. Arch Intern Med. 1986 Oct;146(10):1913-6. PMID 3532983
- [Background] Chang FY, Chou MY. Comparison of pyogenic liver abscesses caused by Klebsiella pneumoniae and non-K. pneumoniae pathogens. J Formos Med Assoc. 1995 May;94(5):232-7. PMID 7613255
- [Background] Yu WL, Chan KS, Ko WC, Lee CC, Chuang YC. Lower prevalence of diabetes mellitus in patients with Klebsiella pneumoniae primary liver abscess caused by isolates of K1/K2 than with non-K1/K2 capsular serotypes. Clin Infect Dis. 2007 Dec 1;45(11):1529-30; author reply 1532-3. doi: 10.1086/523006. No abstract available. PMID 17990242
- [Background] Chung DR, Lee SS, Lee HR, Kim HB, Choi HJ, Eom JS, Kim JS, Choi YH, Lee JS, Chung MH, Kim YS, Lee H, Lee MS, Park CK; Korean Study Group for Liver Abscess. Emerging invasive liver abscess caused by K1 serotype Klebsiella pneumoniae in Korea. J Infect. 2007 Jun;54(6):578-83. doi: 10.1016/j.jinf.2006.11.008. Epub 2006 Dec 18. PMID 17175028
- [Background] Tan YM, Chee SP, Soo KC, Chow P. Ocular manifestations and complications of pyogenic liver abscess. World J Surg. 2004 Jan;28(1):38-42. doi: 10.1007/s00268-003-6963-2. Epub 2003 Nov 14. PMID 14612992
- [Background] Yeoh KG, Yap I, Wong ST, Wee A, Guan R, Kang JY. Tropical liver abscess. Postgrad Med J. 1997 Feb;73(856):89-92. doi: 10.1136/pgmj.73.856.89. PMID 9122104
- [Background] Okano H, Shiraki K, Inoue H, Kawakita T, Yamamoto N, Deguchi M, Sugimoto K, Sakai T, Ohmori S, Murata K, Nakano T. Clinicopathological analysis of liver abscess in Japan. Int J Mol Med. 2002 Nov;10(5):627-30. PMID 12373305
- [Background] Wiwanitkit V. Causative agents of liver abscess in HIV-seropositive patients: a 10-year case series in Thai hospitalized patients. Trop Doct. 2005 Apr;35(2):115-7. doi: 10.1258/0049475054036904. PMID 15970044
- [Background] Lederman ER, Crum NF. Pyogenic liver abscess with a focus on Klebsiella pneumoniae as a primary pathogen: an emerging disease with unique clinical characteristics. Am J Gastroenterol. 2005 Feb;100(2):322-31. doi: 10.1111/j.1572-0241.2005.40310.x. PMID 15667489
- [Background] Nadasy KA, Domiati-Saad R, Tribble MA. Invasive Klebsiella pneumoniae syndrome in North America. Clin Infect Dis. 2007 Aug 1;45(3):e25-8. doi: 10.1086/519424. Epub 2007 Jun 18. PMID 17599300
- [Background] Keynan Y, Karlowsky JA, Walus T, Rubinstein E. Pyogenic liver abscess caused by hypermucoviscous Klebsiella pneumoniae. Scand J Infect Dis. 2007;39(9):828-30. doi: 10.1080/00365540701266763. PMID 17701725
- [Background] Karama EM, Willermain F, Janssens X, Claus M, Van den Wijngaert S, Wang JT, Verougstraete C, Caspers L. Endogenous endophthalmitis complicating Klebsiella pneumoniae liver abscess in Europe: case report. Int Ophthalmol. 2008 Apr;28(2):111-3. doi: 10.1007/s10792-007-9111-4. Epub 2007 Aug 1. PMID 17668150
- [Background] Rahimian J, Wilson T, Oram V, Holzman RS. Pyogenic liver abscess: recent trends in etiology and mortality. Clin Infect Dis. 2004 Dec 1;39(11):1654-9. doi: 10.1086/425616. Epub 2004 Nov 9. PMID 15578367
- [Background] Harris PJ, Laczek JT, Polish RD, Fraser SL. Two cases of Klebsiella pneumoniae primary liver abscesses; an emerging clinical entity among diabetics. Hawaii Med J. 2005 Dec;64(12):306-7, 325. PMID 16438021
- [Background] Yu SC, Ho SS, Lau WY, Yeung DT, Yuen EH, Lee PS, Metreweli C. Treatment of pyogenic liver abscess: prospective randomized comparison of catheter drainage and needle aspiration. Hepatology. 2004 Apr;39(4):932-8. doi: 10.1002/hep.20133. PMID 15057896
- [Background] Wang JH, Liu YC, Lee SS, Yen MY, Chen YS, Wang JH, Wann SR, Lin HH. Primary liver abscess due to Klebsiella pneumoniae in Taiwan. Clin Infect Dis. 1998 Jun;26(6):1434-8. doi: 10.1086/516369. PMID 9636876
- [Background] Chen YW, Chen YS, Lee SS, Yen MY, Wann SR, Lin HH, Huang WK, Liu YC. A pilot study of oral fleroxacin once daily compared with conventional therapy in patients with pyogenic liver abscess. J Microbiol Immunol Infect. 2002 Sep;35(3):179-83. PMID 12380791
- [Background] Zerem E, Hadzic A. Sonographically guided percutaneous catheter drainage versus needle aspiration in the management of pyogenic liver abscess. AJR Am J Roentgenol. 2007 Sep;189(3):W138-42. doi: 10.2214/AJR.07.2173. PMID 17715080
- [Background] Edmiston CE, Krepel CJ, Seabrook GR, Somberg LR, Nakeeb A, Cambria RA, Towne JB. In vitro activities of moxifloxacin against 900 aerobic and anaerobic surgical isolates from patients with intra-abdominal and diabetic foot infections. Antimicrob Agents Chemother. 2004 Mar;48(3):1012-6. doi: 10.1128/AAC.48.3.1012-1016.2004. PMID 14982797
- [Background] Chang SC, Fang CT, Hsueh PR, Chen YC, Luh KT. Klebsiella pneumoniae isolates causing liver abscess in Taiwan. Diagn Microbiol Infect Dis. 2000 Aug;37(4):279-84. doi: 10.1016/s0732-8893(00)00157-7. PMID 10974581
- [Background] Sheng WH, Wang JT, Chen YC, Chang SC, Luh KT. In vitro activity of moxifloxacin against common clinical bacterial isolates in Taiwan. J Microbiol Immunol Infect. 2001 Sep;34(3):178-84. PMID 11605808
- [Background] Cheng HP, Siu LK, Chang FY. Extended-spectrum cephalosporin compared to cefazolin for treatment of Klebsiella pneumoniae-caused liver abscess. Antimicrob Agents Chemother. 2003 Jul;47(7):2088-92. doi: 10.1128/AAC.47.7.2088-2092.2003. PMID 12821451
- [Background] Paterson DL. "Collateral damage" from cephalosporin or quinolone antibiotic therapy. Clin Infect Dis. 2004 May 15;38 Suppl 4:S341-5. doi: 10.1086/382690. PMID 15127367
- [Background] Van Saene JJ, Van Saene HK, Geitz JN, Tarko-Smit NJ, Lerk CF. Quinolones and colonization resistance in human volunteers. Pharm Weekbl Sci. 1986 Feb 21;8(1):67-71. doi: 10.1007/BF01975484. PMID 2938072
- [Background] de Vries-Hospers HG, Welling GW, van der Waaij D. Influence of quinolones on throat- and faecal flora of healthy volunteers. Pharm Weekbl Sci. 1987 Dec 11;9 Suppl:S41-4. doi: 10.1007/BF02075258. PMID 3438150